CLINICAL TRIAL: NCT02699320
Title: Multi-center Clinical Research About Standard Diagnosis and Treatment of Neonate Severe Digestive System Malformation
Brief Title: Intestinal Microbial Dysbiosis in Chinese Infants With Short Bowel Syndrome With Different Complications
Acronym: MSBS
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiang WU, MD., Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-001
Record Dates: First submitted 2016-02-02; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Short Bowel Syndrome; Complications
Keywords: Short bowel syndrome; Intestinal microbiota; immune
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- "Asymptomatic": "Asymptomatic" meaning patients showed well tolerance to parenteral nutrient (PN) administration and there were no complications occurred within two months (n=7);
  Interventions: Other: Complications
- CLABSI: with central catheter-related blood stream infections (CLABSI) meaning patients had fever, increased neutrophils, documented positive catheter blood culture but exclude other source of infection (n=5)
  Interventions: Other: Complications
- PNALD: with parenteral nutrient associated liver disease (PNALD), meaning SBS patients showed elevated liver enzymes and bilirubin (n=14).
  Interventions: Other: Complications
- healthy controls: Seven healthy infants who had added complementary were served as controls (n=7).
  Interventions: Other: Complications

INTERVENTIONS:
Other: Complications — Not involved

SUMMARY:
There are no reports involved the intestinal microbiota from Chinese infants with short bowel syndrome (SBS) under different clinical status. Alterations in the microbiota are closely correlated with the bile acids and short chain fatty acids metabolism as well as the intestinal immunity. A relatively comprehensive profile composed of microbial structure, microbial metabolism products and immune biomarkers in SBS infants may facilitate a better therapy strategy to complications occurred in SBS children.

DETAILED DESCRIPTION:
The investigators totally collected 26 fecal samples from 18 infants diagnosed with SBS during parenteral nutrition administration, and these samples were divided into three groups according to complications of enrolled patients at sampling time: asymptomatic group, central catheter-related blood stream infections group and liver injury group. 7 healthy infants with supplementary food were enrolled as control. Fecal microbiota, sIgA and calprotectin, bile acids and short chain fatty acids were also detected by 16S ribosomal ribonucleic acid (rRNA) gene sequencing, enzyme-linked immunosorbent assay and liquid/gas chromatography.

ELIGIBILITY:
Inclusion Criteria:

* Infants with short bowel syndrome

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 18 infants diagnosed with SBS were enrolled from Digestion and Nutrition Division at Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Microbial structure in SBS infants | up to 4 months
  Fecal microbiota were detected by 16S rRNA gene sequencing.

SECONDARY OUTCOMES:
Metabolism products in SBS infants | up to 4 months
  Bile acids and short chain fatty acids were detected by liquid/gas chromatography.
Immune biomarkers in SBS infants | up to 4 months
  Secretary IgA and calprotectin were detected by enzyme-linked immunosorbent assay.

CONTACTS AND LOCATIONS:
Overall Officials: Guangyu Chen, PhD, Principal Investigator — Shanghai Municipal Science and Technology Commission
Locations (1):
- Ethics Committee of Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vanderhoof JA, Langnas AN. Short-bowel syndrome in children and adults. Gastroenterology. 1997 Nov;113(5):1767-78. doi: 10.1053/gast.1997.v113.pm9352883.
- [Result] Wales PW, de Silva N, Kim J, Lecce L, To T, Moore A. Neonatal short bowel syndrome: population-based estimates of incidence and mortality rates. J Pediatr Surg. 2004 May;39(5):690-5. doi: 10.1016/j.jpedsurg.2004.01.036. PMID 15137001
- [Result] Howard L, Ashley C. Management of complications in patients receiving home parenteral nutrition. Gastroenterology. 2003 May;124(6):1651-61. doi: 10.1016/s0016-5085(03)00326-3. PMID 12761723
- [Result] Bull MJ, Plummer NT. Part 1: The Human Gut Microbiome in Health and Disease. Integr Med (Encinitas). 2014 Dec;13(6):17-22. PMID 26770121
- [Result] Caldarini MI, Pons S, D'Agostino D, DePaula JA, Greco G, Negri G, Ascione A, Bustos D. Abnormal fecal flora in a patient with short bowel syndrome. An in vitro study on effect of pH on D-lactic acid production. Dig Dis Sci. 1996 Aug;41(8):1649-52. doi: 10.1007/BF02087915. PMID 8769294
- [Result] Sondheimer JM, Asturias E, Cadnapaphornchai M. Infection and cholestasis in neonates with intestinal resection and long-term parenteral nutrition. J Pediatr Gastroenterol Nutr. 1998 Aug;27(2):131-7. doi: 10.1097/00005176-199808000-00001. PMID 9702641
- [Result] Winter SE, Baumler AJ. Dysbiosis in the inflamed intestine: chance favors the prepared microbe. Gut Microbes. 2014 Jan-Feb;5(1):71-3. doi: 10.4161/gmic.27129. Epub 2014 Jan 29. PMID 24637596
- [Result] Halmos T, Suba I. [Physiological patterns of intestinal microbiota. The role of dysbacteriosis in obesity, insulin resistance, diabetes and metabolic syndrome]. Orv Hetil. 2016 Jan 3;157(1):13-22. doi: 10.1556/650.2015.30296. Hungarian. PMID 26708682
- [Result] Furtado Ede C, Marchini JS, Fonseca CK, Coelho PS, Menegueti MG, Auxiliadora-Martins M, Basile-Filho A, Suen VM. Cyclic parenteral nutrition does not change the intestinal microbiota in patients with short bowel syndrome. Acta Cir Bras. 2013;28 Suppl 1:26-32. doi: 10.1590/s0102-86502013001300006. PMID 23381820
- [Result] Joly F, Mayeur C, Bruneau A, Noordine ML, Meylheuc T, Langella P, Messing B, Duee PH, Cherbuy C, Thomas M. Drastic changes in fecal and mucosa-associated microbiota in adult patients with short bowel syndrome. Biochimie. 2010 Jul;92(7):753-61. doi: 10.1016/j.biochi.2010.02.015. Epub 2010 Feb 19. PMID 20172013
- [Result] Engstrand Lilja H, Wefer H, Nystrom N, Finkel Y, Engstrand L. Intestinal dysbiosis in children with short bowel syndrome is associated with impaired outcome. Microbiome. 2015 May 4;3:18. doi: 10.1186/s40168-015-0084-7. eCollection 2015. PMID 25941569
- [Result] Davidovics ZH, Carter BA, Luna RA, Hollister EB, Shulman RJ, Versalovic J. The Fecal Microbiome in Pediatric Patients With Short Bowel Syndrome. JPEN J Parenter Enteral Nutr. 2016 Nov;40(8):1106-1113. doi: 10.1177/0148607115591216. Epub 2015 Jun 9. PMID 26059898
- [Result] Bharadwaj S, Gohel T, Deen OJ, DeChicco R, Shatnawei A. Fish oil-based lipid emulsion: current updates on a promising novel therapy for the management of parenteral nutrition-associated liver disease. Gastroenterol Rep (Oxf). 2015 May;3(2):110-4. doi: 10.1093/gastro/gov011. Epub 2015 Apr 8. PMID 25858884
- [Result] Raphael BP, Mitchell PD, Finkton D, Jiang H, Jaksic T, Duggan C. Necrotizing Enterocolitis and Central Line Associated Blood Stream Infection Are Predictors of Growth Outcomes in Infants with Short Bowel Syndrome. J Pediatr. 2015 Jul;167(1):35-40.e1. doi: 10.1016/j.jpeds.2015.02.053. Epub 2015 Apr 1. PMID 25841540
- [Result] Greenberg RG, Moran C, Ulshen M, Smith PB, Benjamin DK Jr, Cohen-Wolkowiez M. Outcomes of catheter-associated infections in pediatric patients with short bowel syndrome. J Pediatr Gastroenterol Nutr. 2010 Apr;50(4):460-2. doi: 10.1097/MPG.0b013e3181b99d07. PMID 20179637
- [Result] Kurkchubasche AG, Smith SD, Rowe MI. Catheter sepsis in short-bowel syndrome. Arch Surg. 1992 Jan;127(1):21-4; discussion 24-5. doi: 10.1001/archsurg.1992.01420010027004. PMID 1734846
- [Result] Sayin SI, Wahlstrom A, Felin J, Jantti S, Marschall HU, Bamberg K, Angelin B, Hyotylainen T, Oresic M, Backhed F. Gut microbiota regulates bile acid metabolism by reducing the levels of tauro-beta-muricholic acid, a naturally occurring FXR antagonist. Cell Metab. 2013 Feb 5;17(2):225-35. doi: 10.1016/j.cmet.2013.01.003. PMID 23395169
- [Result] Pereira-Fantini PM, Lapthorne S, Joyce SA, Dellios NL, Wilson G, Fouhy F, Thomas SL, Scurr M, Hill C, Gahan CG, Cotter PD, Fuller PJ, Hardikar W, Bines JE. Altered FXR signalling is associated with bile acid dysmetabolism in short bowel syndrome-associated liver disease. J Hepatol. 2014 Nov;61(5):1115-25. doi: 10.1016/j.jhep.2014.06.025. Epub 2014 Jul 3. PMID 24999016
- [Result] Amato KR, Yeoman CJ, Kent A, Righini N, Carbonero F, Estrada A, Gaskins HR, Stumpf RM, Yildirim S, Torralba M, Gillis M, Wilson BA, Nelson KE, White BA, Leigh SR. Habitat degradation impacts black howler monkey (Alouatta pigra) gastrointestinal microbiomes. ISME J. 2013 Jul;7(7):1344-53. doi: 10.1038/ismej.2013.16. Epub 2013 Mar 14. PMID 23486247
- [Result] Treem WR, Ahsan N, Shoup M, Hyams JS. Fecal short-chain fatty acids in children with inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 1994 Feb;18(2):159-64. doi: 10.1097/00005176-199402000-00007. PMID 8014762
- [Result] Michon AL, Aujoulat F, Roudiere L, Soulier O, Zorgniotti I, Jumas-Bilak E, Marchandin H. Intragenomic and intraspecific heterogeneity in rrs may surpass interspecific variability in a natural population of Veillonella. Microbiology (Reading). 2010 Jul;156(Pt 7):2080-2091. doi: 10.1099/mic.0.038224-0. Epub 2010 Apr 22. PMID 20413553
- [Result] Delwiche EA, Pestka JJ, Tortorello ML. The veillonellae: gram-negative cocci with a unique physiology. Annu Rev Microbiol. 1985;39:175-93. doi: 10.1146/annurev.mi.39.100185.001135. No abstract available. PMID 3904599
- [Result] Bhatti MA, Frank MO. Veillonella parvula meningitis: case report and review of Veillonella infections. Clin Infect Dis. 2000 Sep;31(3):839-40. doi: 10.1086/314046. PMID 11017846
- [Result] Chichlowski M, Hale LP. Bacterial-mucosal interactions in inflammatory bowel disease: an alliance gone bad. Am J Physiol Gastrointest Liver Physiol. 2008 Dec;295(6):G1139-49. doi: 10.1152/ajpgi.90516.2008. Epub 2008 Oct 16. PMID 18927210
- [Result] Demehri FR, Barrett M, Ralls MW, Miyasaka EA, Feng Y, Teitelbaum DH. Intestinal epithelial cell apoptosis and loss of barrier function in the setting of altered microbiota with enteral nutrient deprivation. Front Cell Infect Microbiol. 2013 Dec 23;3:105. doi: 10.3389/fcimb.2013.00105. eCollection 2013. PMID 24392360
- [Result] Nolan JP. Intestinal endotoxins as mediators of hepatic injury--an idea whose time has come again. Hepatology. 1989 Nov;10(5):887-91. doi: 10.1002/hep.1840100523. No abstract available. PMID 2680869
- [Result] Guarner F, Wallace JL, MacNaughton WK, Ibbotson GC, Arroyo V, Rodes J. Endotoxin-induced ascites formation in the rat: partial mediation by platelet-activating factor. Hepatology. 1989 Nov;10(5):788-94. doi: 10.1002/hep.1840100507. PMID 2807157